CLINICAL TRIAL: NCT05578014
Title: Survey on Change Temperature of Skin Surface at the Acupuncture Site, the Neck and the Face When Using Tonifying Acupuncture Manipulations or Dispersing Acupuncture Manipulations at Dazhui in Healthy Volunteers: a Pilot Study
Brief Title: Change Temperature of Skin Surface at the Acupuncture Site, the Neck and the Face When Using Tonifying Acupuncture Manipulations or Dispersing Acupuncture Manipulations at Dazhui in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bui Pham Minh Man (Other)
Responsible Party: Sponsor-Investigator, Bui Pham Minh Man, Medical Doctor, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 678/HDDD-DHYD
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers
Keywords: Acupuncture Manipulations; Tonifying Acupuncture Manipulations; Dispersing Acupuncture Manipulations
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: A pilot study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group STD (Experimental): 19 participant received sham acupuncture at EX-B2 T3 point in right side or acupuncture with tonyfying or dispersing manipulations at Dazhui point, corresponding to 3 times of acupuncture in 14 days, each time is 7 days aparts. In each time, temperature of skin surface at the acupuncture site, the neck and the face will be recorded.
  Procedure/Surgery: Acupuncture with disposable acupuncture needles (the size of 0.30 x 25 mm) at EX-B2 T3 point in right side as sham acupoint in the first trial phase. We used the same type of acupuncture needles as aboved to acupuncture at Dazhui with tonifying manipulations in the second trial phase and with dispersing manipulatiuons in the third trial phase.
  Interventions: Procedure: Acupuncture
- Group TDS (Experimental): 19 participant received acupuncture with tonyfying or dispersing manipulations at Dazhui or sham acupuncture at EX-B2 T3 point in right side, corresponding to 3 times of acupuncture in 14 days, each time is 7 days aparts. In each time, temperature of skin surface at the acupuncture site, the neck and the face will be recorded.
  Procedure/Surgery: Acupuncture with disposable acupuncture needles (the size of 0.30 x 25 mm) at Dazhui with tonifying manipulations in the first trial phase and with dispersing manipulatiuons in the second trial phase. We used the same type of acupuncture needles as aboved to acupuncture at EX-B2 T3 point in right side as sham acupoint in the third trial phase.
  Interventions: Procedure: Acupuncture
- Group DST (Experimental): 19 participant received acupuncture with tonyfying or dispersing manipulations at Dazhui or sham acupuncture at EX-B2 T3 point in right side, corresponding to 3 times of acupuncture in 14 days, each time is 7 days aparts. In each time, temperature of skin surface at the acupuncture site, the neck and the face will be recorded.
  Procedure/Surgery: Acupuncture with disposable acupuncture needles (the size of 0.30 x 25 mm) at Dazhui with tonifying manipulations in the first trial phase and with dispersing manipulatiuons in the second trial phase. We used the same type of acupuncture needles as aboved to acupuncture at EX-B2 T3 point in right side as sham acupoint in the third trial phase.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — To conduct this intervention, we used disposable acupuncture needles with the size of 0.30 x 25 mm to acupuncture the sham acupoint (EX-B2 T3 point) or Dazhui point.

SUMMARY:
Acupuncture is a treatment method since ancient times and it has been recognized as an international treatment method by the World Health Organization. Although the structure and physiological effects of acupoints have been extensively studied, they have not been fully elucidated. A lot of studies on physiological effects of acupoints on the 12 main merdians have been published, but acupoints outside the meridians or acupoints on the eight extraordinary vessels have not been noticed. In particular, the Dazhui is one of the acupoints on the Du Merdian that is often used clinically. In the other side, several researches have shown that using different acupuncture manipulations can achieve different therapeutic effects. In our study, we want to determinate and compare the change temperature of skin surface at the acupuncture site, the neck and the face when using tonifying acupuncture manipulations or dispersing acupuncture manipulations at Dazhui in healthy volunteers.

DETAILED DESCRIPTION:
Participants and Methods: A pilot study is conducted by comparing the change in skin surface temperature before and after using sham or tonifying or dispersing acupuncture manipulations at EX-B2 T3 in right side and Dazhui in heatlhy volunteers. A total of 57 participants will be randomly divided into 3 groups (group STD, group TDS and group DST). Each group has 19 participants and undergo 3 trial phases, corresponding to 3 times of acupuncture in 14 days, each time is 7 days apart. For group STD, the first trial phase: participants received acupuncture at EX-B2 T3 point in right side as sham acupuncture; the second trial phase: participants received acupuncture with tonifying manipulations at Dazhui point and tonifying manipulations was replaced by dispersing ones in the third trial phase. For group TDS, the first trial phase: participants received acupuncture with tonifying manipulations at Dazhui point; the second trial phase: participants received acupuncture with dispersing manipulations at Dazhui point and participants received acupuncture at EX-B2 T3 point in right side as sham acupuncture in the third trial phase. Similarly, for group DST, the first trial phase: participants received acupuncture with dispersing manipulations at Dazhui point; the second trial phase: participants received acupuncture at EX-B2 T3 point in right side as sham acupuncture and sham acupuncture was replaced byacupuncture with tonifying manipulations at Dazhui in the third trial phase. The primary outcome was the change temperature of skin surface at the acupuncture site, the neck and the face when using tonifying or dispersing acupuncture manipulations at Dazhui point. This trial will be performed as a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, regardless of gender or profession
* Age between enough 18 and 30 years old.
* BMI: 18.5 - 23 kg/m2
* Mental alertness, good contact, cooperation with researchers.
* DASS 21 score within normal limits.
* Have no disease which change the body temperature, like hyperthyroidism, hypothyroidism.
* Vital sign within normal limits:

  * Heart rates from from 60 to 100 beats/minute.
  * Systolic blood pressure between 90 and 139 mmHg.
  * Diastolic blood pressure between 60 and 89 mmHg.
  * Body temperature: 36.59 ± 0.43 0C.
  * SpO2 from 95 to 99%.
* Volunteers who agree to participate and sign the Informed Consent Form, following a detailed explanation of clinical trials.
* Not currently participating in other intervention studies.
* Have no acupuncture experience yet.

Exclusion Criteria:

* Having an inflammatory injury in the site of the skin to be investigated.
* Using heat therapy, for example massage, cupping therapy, acupuncture in the site of the skin to be investigated within 24h.
* Applying chemical or pharmaceutical products to the site of the skin to be survey before conducting the study.
* Other diseases that could affect or interfere with outcomes, including common cold or flu.
* Curently having neck-pain or having skin diseases, for example: tinea versicolor, eczema in the site of the skin to be investigated.
* Taking stimulant (alcohol, beer, coffee, tobacco) within 24h.
* Staying up at night or having insomnia before the day of the study.
* Playing sport within 2h.
* Pregnant woman or breastfeeding woman or woman in period.
* Currently using certain drugs which dilate blood vessels and drop in blood pressure.
* Anxiety, depression, stress before conducting the study with DASS 21 score < 15.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change temperature of skin surface at at the acupuncture site, the neck and the face when using tonifying acupuncture manipulations at Dazhui | During procedure
Change temperature of skin surface at at the acupuncture site, the neck and the face when using dispersing acupuncture manipulations at Dazhui | During procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Traditional medicine - University of Medicine and Pharmacy of Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Demographic characteristic and outcome data will be shared
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- See also: World Health Organization. Acupuncture : review and analysis of reports on controlled clinical trials. World Health Organization; 2014.May 16, 2022. — https://chiro.org/acupuncture/FULL/Acupuncture_WHO_2003.pdf
- See also: Z. Lu, H. Dong, Q. Wang, et al. Perioperative acupuncture modulation: more than anaesthesia. doi:10.1093/bja/aev227British Journal of Anaesthesia.2015;115(2):183-193. — https://pubmed.ncbi.nlm.nih.gov/26170347/
- See also: Jia-Min Yang, Xiao-Yu Shen, Ling Zhang, et al. The Effect of Acupuncture to SP6 on Skin Temperature Changes of SP6 and SP10: An Observation of "Deqi". Evidence-Based Complementary and Alternative Medicine. 2014;2014: 595963. Doi: 10.1155/2014/595963 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3934096/
- See also: Ali Mohammadi, Liang-Xiao Ma, Yang Yang, et al. Immediate Analgesic Effect of Perpendicular Needling or Transverse Needling at SP6 in Primary Dysmenorrhea: A Pilot Study. Medical Acupuncture. 2019;31(4): 207-217. Doi:10.1089/acu.2019.1362 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6709727/
- See also: Weihui Li, Andrew Ahn. Effect of Acupuncture Manipulations at LI4 or LI11 on Blood Flow and Skin Temperature. Journal of Acupuncture & Meridian Studies. 2016;9(3):128-133. doi:10.1016/j.jams.2015.08.005 — https://pubmed.ncbi.nlm.nih.gov/23476709/